# Hualien Tzu Chi Hospital The Application for In-Hospital Medical Technology Research Project

Application Number:

## 1.Basic Information

| | ■Individual Re | esearch Project: | The project | leader is a senior staff r | nember of the |
|---|---|---|---|---|---|
| | hospital. | | | | |
| | Experimental | Research (Up to | o 800,000 N | ITD | |
| | □Non-Experin | nental Research ( | (Up to 400,0 | 000 NTD) | |
| | ☐Holistic Care | Departmental P | roject (Up t | o 800,000 NTD) (Only | department heads |
| Project Category | are eligible to | apply) | | | |
| (Select one) | □New Staff Re | esearch Project ( | Up to 200,0 | 00 NTD) | |
| | University-H | ospital Collabora | ative Resear | rch Project (Up to 400,0 | 000 NTD) |
| | ☐Ministry of S | cience and Tech | nology Trai | nsfer to Hospital Project | t (Up to 800,000 |
| | NTD) | | | | |
| | Medical Education Research Project (Up to 400,000 NTD) | | | | |
| Personnel Category | <b>-</b> D1 :: | | | | |
| (Select one) | Physician Non-Physician | | | | |
| Project Title | | • • | | pervigilance in disorder<br>d cognitive-behavioral | _ |
| Name of the Project | Wei-Yi Lei | Title/Position | Attending | Applying | Gastroenterology |
| Leader | wei- i i Lei | Title/Position | Physician | Department/Division | Department |
| Project Execution Period | From January 1 | , 2024 to Decem | ber 31, 202 | 5 | |
| | Basic Resear | ch Applied F | Research | Technology Develop | oment |
| | (Note: Those w | ho select Applie | d Research | and Technology Develo | pment must also |
| | select the category of Innovation R&D.) | | | | |
| Research Nature | Innovation R&D Classification: ■(1) Clinical Research | | | | |
| and Classification | (2) Translational Research (3) Medical Engineering and Materials | | | | |
| | (4) Informatio (5) Medical Assistance Operations (6) Others, please specify | | | | |
| | o | | | | |
| | Holistic Care C | lassification: | | | |
| Holistic Care (Please refer to the | (1) Patient-Cent | tered ( Physica | al, 🗌 Psych | ological, Environme | ental, Spiritual) |
| term description, | (2) Health Ed | ucation ( Be | havior Cha | nge, Health Prom | otion, Disease |
| multiple selections | | Early Diagnosis, | ☐ Early Tı | reatment) | |
| are allowed) | (2) Others places specify | | | | |

| Has this in-house proj | ect applied for the 2023 Ministry of Science and Technology's Special Research |
|---|---|
| Program? | |
| ■ No □ Yes. | |
| Has any government a | gency subsidy for research projects been applied for this year? |
| ☐ No ■ Yes, a total | of 1 projects. |
| A total of 1 in-ho | use research projects have been applied for this year as the principal investigator |
| (jointly hosted project | s are not included). |
| The priority of this pro | oject is 1. |
| Has this project applie | od for: |
| ☐ No need | |
| ■ Human Experimen | ts / Human Samples (including human embryos/human embryonic stem cells) |
| ☐ Animal Experimen | ts |
| ☐ Biosafety (includin | g recombinant DNA experiments/genetically modified organism field trials/Level 2 or |
| higher infectious biolo | ogical materials) |
| [Please check the ap | plicable items |
| | Name: Lei Wei-Yi |
| Project Contact | Phone: (Office) (03) 8561825-13224 (Home) 0970-339629 |
| Person | E-Mail: aquarious@seed.net.tw |

2. **Application for Subsidy Funding** (The budget allocation will be included in the review and evaluation criteria, please do not inflate the figures.)

Based on the actual needs of the research project, the following items can be applied for subsidy funding:

- For individual research projects:
  - o Experimental research: Maximum of 800,000 NTD
  - o Non-experimental research: Maximum of 400,000 NTD
- For new personnel research projects: The total research funding is limited to 200,000 NTD.
- For collaborative research projects between schools and institutions: The total research funding is limited to 400,000 NTD.
- For holistic care department projects: The maximum funding is 800,000 NTD.
- For Ministry of Science and Technology transferred in-house projects: The maximum funding is 800,000 NTD.

| Subsidy Items | | Requested Amount |
|---|---|---|
| Administrative<br>Expenses | 1. Research<br>Personnel Costs | 480,000 NTD |
| | 2. Experimental Animal Costs | 0 NTD |
| | 3. Consumables,<br>Materials, Books,<br>and Miscellaneous<br>Expenses | 160,000 NTD |
| Research Equipment Costs | | 0 NTD |
| Total Amount | | 640,000 NTD |

## 3. Equipment Configuration

The names of the main instruments required for this project, their placement locations, and the signature of the responsible person consenting to their use.

| Instrument Name | Installation Location (Department) | Signature and Seal of the Department Head Approving the Use of the Instrument |
|---|---|---|

## 4. Personnel Involved in the Project

## (1) Principal Research Personnel

| | | T | 1 |
|---|---|---|---|
| Category (Principal Investigator, Co-Principal Investigator, Collaborating Principal Investigator, Research Assistant, etc.) | Name | Current Position | Specific Job Role, Tasks, and Scope of Work in this Research Project |
| Principal<br>Investigator | Lei Wei-Yi | Attending Physician, Gastroenterology | Research project planning and participant recruitment, progress monitoring, data statistical analysis, and report writing. |
| Co-Principal<br>Investigator | Chen Jian-<br>Lin | Director of Gastroenterology<br>Department | Project progress supervision, project planning discussions, participant recruitment, and data analysis. |
| Co-Principal<br>Investigator | Weng Ming-<br>Wen | Attending Physician, Gastroenterology | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Yi Zhi-Xun | Attending Physician, Gastroenterology | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Liu Zuo-Cai | Director of the Digestive<br>Function Testing Department | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Hong Rui-<br>Sheng | Attending Physician,<br>Gastroenterology | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Wang Jun-<br>Wei | Attending Physician, Gastroenterology Department, Kaohsiung Medical University Hospital | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Liang Shu-<br>Wei | Attending Physician, Gastroenterology Department, Chung Shan Medical University Hospital | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Wang Wen-<br>Hui | Director of Gastroenterology<br>Department, E-Da Hospital | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Hsieh Ming-<br>Tsung | Attending Physician, Gastroenterology Department, National Cheng Kung University Hospital | Research project participant recruitment and actual case handling. |
| Co-Principal<br>Investigator | Lin Yi-Mei | Professor, Department of<br>Psychology, Kaohsiung<br>Medical University | Cognitive Behavioral Therapy coordination and data analysis. |
| Co-Principal<br>Investigator | Lin Hui-Min | Dietitian, Clinical Nutrition Division, Department of Nutrition | Developing nutrition education materials and arranging the nutrition consultation process. |

| Research<br>Personnel | Lin Pei-Yun | Psychotherapist, Yuli Hospital | Conducting Cognitive Behavioral Therapy. |
|---|---|---|---|
| Research<br>Personnel | Hsu Ssu-Ting | Counseling Psychologist,<br>Secret Garden Counseling<br>Center | Conducting Cognitive Behavioral Therapy. |
| Research<br>Personnel | ISu Zhen- | Dietitian, Clinical Nutrition Division, Department of Nutrition | Conducting nutrition counseling and education. |
| Research<br>Assistant | Huang Chun-<br>Hsiang | lResearch Assistant | Survey administration, data collection, organization and analysis, and handling administrative tasks. |

<sup>\*</sup>If there are insufficient fields, please copy them as needed.

## (2) Research projects that the principal investigator, co-principal investigator, and coresearchers have participated in during the past three years.

| Name | Project Name | Role and<br>Responsibilities in the<br>Project | Start and<br>End Date | Funding<br>Agency |
|---|---|---|---|---|
| Lei Wei-<br>Yi | Exploring the roles and interrelationships of esophageal hypersensitivity, psychological distress, and functional gastrointestinal disorders in the pathophysiological mechanisms of esophageal symptoms in patients. | Principal Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Exploring the pathophysiological mechanisms and treatment strategies of gastroesophageal reflux disease (GERD) through the distribution of afferent nerves, esophageal motility, and pharmacological regulation. | Principal Investigator | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Lei Wei-<br>Yi | Exploring the effects of opioid analysesics on the pathophysiological mechanisms of esophageal contraction and reflux characteristics, as well as their clinical applications. | Principal Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | The efficacy of Jingsi Herbal Concentrate on long COVID symptoms—gut-brain axis dysregulation and related physical and mental symptoms: A randomized double-blind clinical trial. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Foundation |
| Lei Wei-<br>Yi | Exploring the interaction between upper gastric belching, physical and mental symptoms, and esophageal acid reflux: Clinical applications for optimizing the treatment of gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Using high-resolution pharyngeal function testing to analyze the pharyngeal swallowing physiology and dynamics in patients with ineffective esophageal motility. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Exploring the efficacy and physiological changes of anti-reflux mucosal ablation in proton pump inhibitor (PPI)-dependent gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |

| | ersion Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| Lei Wei-<br>Yi | Exploring the sensitivity to capsaicin, motility sensation function, and the physiological features of reflux in the esophagus: Clinical impact and treatment guidelines for esophageal dysfunction and gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Lei Wei-<br>Yi | Exploring the pathophysiological mechanisms of gastroesophageal reflux disease (GERD) through esophageal reflux clearance capacity, mucosal integrity, and psychosocial characteristics, and establishing a basis for precise diagnosis and treatment. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | The application of high-resolution impedance pharyngeal function testing and the Sydney Swallowing Questionnaire in oropharyngeal dysphagia and voice disorders. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | The application of artificial intelligence in high-<br>resolution esophageal function testing: A study on<br>unsupervised computational models based on deep<br>learning. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Application of supervised learning artificial intelligence in analyzing 24-hour esophageal pH-impedance monitoring: Technological efficacy and clinical applications in diagnosing gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Exploring the clinical characteristics and the impact of gut microbiota in patients with metabolic-associated fatty liver disease under dietary and exercise regulation. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | The efficacy of Jingsi Herbal Drink on the physical and mental symptoms of functional dyspepsia: A randomized double-blind clinical trial. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Foundation |
| Lei Wei-<br>Yi | Exploring the pathophysiological role of esophageal mucosal afferent nerve distribution in gastroesophageal reflux disease (GERD) with concurrent esophageal motility dysfunction. | Principal Investigator | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Lei Wei-<br>Yi | Exploring the pathophysiological impact of esophageal contraction, mucosal integrity, and acid sensitivity on gastroesophageal reflux disease (GERD) and the basis for treatment strategies. | Co-Principal<br>Investigator | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Lei Wei-<br>Yi | Exploring the role of esophageal microbiota in gastroesophageal reflux disease (GERD) through novel impedance parameters, clinical subtypes, and hypersensitivity. | Co-Principal<br>Investigator | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Exploring the interrelationship and pathogenic mechanisms of esophageal acid sensitivity, secondary esophageal contractions, and subtypes of gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei Wei-<br>Yi | Exploring the clinical application of high-<br>resolution impedance pharyngeal function testing<br>in oropharyngeal dysphagia and drug response. | Co-Principal<br>Investigator | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Chen<br>Jian-Lin | The efficacy of Jingsi Herbal Concentrate on long COVID symptoms—gut-brain axis dysregulation | Principal Investigator | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Foundation |

| v | ersion Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| | and related physical and mental symptoms: A | | | |
| | randomized double-blind clinical trial. | | | |
| Chen | Exploring the interaction between upper gastric | | | |
| Jian-Lin | belching, physical and mental symptoms, and | | 2023/01/01~ | Hualien Tzu |
| | esophageal acid reflux: Clinical applications for | Principal Investigator | 2023/01/01~ | |
| | optimizing the treatment of gastroesophageal | | 2023/12/31 | Chi Hospital |
| | reflux disease (GERD). | | | |
| Chen | Exploring the relationship between esophageal | | | |
| Jian-Lin | capsaicin sensitivity, motility sensation function, | | | Ministry of |
| | and the physiological characteristics of reflux: | Duin ain al Investigatan | 2023/8/1~ | Science and |
| | Clinical impacts and treatment guidelines for | Principal Investigator | 2026/07/31 | Technology |
| | esophageal dysfunction and gastroesophageal | | | (MOST) |
| | reflux disease (GERD). | | | • |
| Chen | The efficacy of Jingsi Herbal Drink on the physical | | 2022/1/1 | Tzu Chi |
| Jian-Lin | and mental symptoms of functional dyspepsia: A | Principal Investigator | 2022/1/1~ | Medical |
| | randomized double-blind clinical trial. | 1 C | 2022/12/31 | Foundation |
| Chen | Exploring the pathophysiological mechanisms of | | | |
| Jian-Lin | gastroesophageal reflux disease (GERD) through | | | |
| | esophageal reflux clearance capacity, mucosal | | 2022/1/1~ | Hualien Tzu |
| | integrity, and psychosocial characteristics, and | Principal Investigator | 2022/12/31 | Chi Hospital |
| | establishing a basis for precise diagnosis and | | | 1 |
| | treatment. | | | |
| Chen | Exploring the pathophysiological mechanisms and | | | |
| Jian-Lin | interrelationships of esophageal hypersensitivity, | G D: : 1 | 2022/01/01 | |
| | psychological distress, and functional | Co-Principal | 2023/01/01~ | Hualien Tzu |
| | gastrointestinal disorders in patients with | Investigator | 2023/12/31 | Chi Hospital |
| | esophageal symptoms. | | | |
| Chen | Exploring the efficacy and physiological changes | | | |
| Jian-Lin | of anti-reflux mucosal ablation in proton pump | Co-Principal | 2023/01/01~ | Hualien Tzu |
| | inhibitor (PPI)-dependent gastroesophageal reflux | Investigator | 2023/12/31 | Chi Hospital |
| | disease (GERD). | | | |
| Chen | Using high-resolution pharyngeal function testing | | | |
| Jian-Lin | to analyze the pharyngeal swallowing physiology | Co-Principal | 2023/01/01~ | Hualien Tzu |
| 2111 | and dynamics in patients with ineffective | Investigator | 2023/12/31 | Chi Hospital |
| | esophageal motility. | 111 / <b>2</b> 211 <b>8</b> 11-21 | 2020, 12, 61 | om morphum |
| Chen | Exploring the pathophysiological mechanisms of | | | Ministry of |
| Jian-Lin | laryngopharyngeal reflux: Clinical applications of | Co-Principal | 2022/8/1~ | Science and |
| 2111 | artificial intelligence-assisted, precision | Investigator | 2025/07/31 | Technology |
| | diagnostics, and personalized treatment strategies. | C | | (MOST) |
| Chen | Exploring the pathophysiological mechanisms and | | | |
| Jian-Lin | treatment strategies of gastroesophageal reflux | | 2022/0/1 | Ministry of |
| | disease (GERD) through the distribution of | Co-Principal | 2022/8/1~ | Science and |
| | afferent nerves, esophageal motility, and | Investigator | 2025/07/31 | Technology |
| | pharmacological regulation. | | | (MOST) |
| Chen | Exploring the effects of opioid analgesics on the | | | |
| Jian-Lin | pathophysiological mechanisms of esophageal | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | contraction and reflux characteristics, as well as | Investigator | 2022/12/31 | Chi Hospital |
| | their clinical applications. | 2 | | 1 |
| Chen | Application of supervised learning artificial | | | |
| Jian-Lin | intelligence in analyzing 24-hour esophageal pH- | G D: 1 | 2022/1/1 | II 1' T |
| | impedance monitoring: Technological efficacy and | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | clinical applications in diagnosing | Investigator | 2022/12/31 | Chi Hospital |
| | gastroesophageal reflux disease (GERD). | | | |
| | 1 U (). | | l . | |

| | /ersion Date : (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| Chen<br>Jian-Lin | The application of high-resolution impedance pharyngeal function testing and the Sydney | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | Swallowing Questionnaire in oropharyngeal dysphagia and voice disorders. | Investigator | 2022/12/31 | Chi Hospital |
| Chen | The application of artificial intelligence in high- | | | |
| Jian-Lin | resolution esophageal function testing: A study on | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | unsupervised computational models based on deep learning. | Investigator | 2022/12/31 | Chi Hospital |
| Chen | Exploring the clinical characteristics and the impact | C D: 1 | 2022/1/1 | II 1' T |
| Jian-Lin | of gut microbiota in patients with metabolic- | Co-Principal | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| | associated fatty liver disease under dietary and exercise regulation. | Investigator | 2022/12/31 | Cili Hospitai |
| Chen | Exploring the role of esophageal microbiota in | | | |
| Jian-Lin | gastroesophageal reflux disease (GERD) through | Principal Investigator | 2021/1/1~ | Hualien Tzu |
| | novel impedance parameters, clinical subtypes, and hypersensitivity. | Timelput mvestigator | 2021/12/31 | Chi Hospital |
| Chen | Exploring the interrelationship and pathogenic | a <b>n</b> | 0001/1/1 | ** 1. = |
| Jian-Lin | mechanisms of esophageal acid sensitivity, | Co-Principal | 2021/1/1~ | Hualien Tzu |
| | secondary esophageal contractions, and subtypes of gastroesophageal reflux disease (GERD). | Investigator | 2021/12/31 | Chi Hospital |
| Chen | Exploring the clinical application of high- | Co. Dain aireal | 2021/1/1 | Hastina Ten |
| Jian-Lin | resolution impedance pharyngeal function testing | Co-Principal<br>Investigator | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| | in oropharyngeal dysphagia and drug response. | | 2021/12/31 | |
| Chen | Exploring the pathophysiological role of | C. D 1 | 2020/0/1 | Ministry of |
| Jian-Lin | esophageal mucosal afferent nerve distribution in gastroesophageal reflux disease (GERD) with | Co-Principal<br>Investigator | 2020/8/1~<br>2022/07/31 | Science and Technology |
| Chen | concurrent esophageal motility dysfunction. | | | (MOST) |
| Jian-Lin | Improving the diagnosis of laryngopharyngeal reflux through the proximal esophageal nighttime | | | Ministry of |
| | average baseline mucosal impedance values and | Co-Principal | 2020/8/1~ | Science and |
| | establishing the indications for proton pump inhibitor therapy. | Investigator | 2022/07/31 | Technology (MOST) |
| Chen | Exploring the pathophysiological impacts of | | | Ministry of |
| Jian-Lin | esophageal contraction, mucosal integrity, and acid | | 2020/8/1~ | Ministry of Science and |
| | sensitivity on gastroesophageal reflux disease | Principal Investigator | 2023/07/31 | Technology |
| | (GERD), and establishing treatment strategies based on these factors. | | | (MOST) |
| Weng | Exploring the efficacy and physiological changes | | | |
| Ming- | of anti-reflux mucosal ablation in proton pump | Dringing! Investigate | 2023/01/01~ | Hualien Tzu |
| Wen | inhibitor (PPI)-dependent gastroesophageal reflux disease (GERD). | Principal Investigator | 2023/12/31 | Chi Hospital |
| Weng | Exploring the pathophysiological mechanisms of | | | Ministry of |
| Ming- | laryngopharyngeal reflux: Clinical applications of | Principal Investigator | 2022/8/1~ | Science and |
| Wen | artificial intelligence-assisted precision diagnostics and personalized treatment strategies. | Timelpar mivestigator | 2025/07/31 | Technology (MOST) |
| Weng | Using supervised learning artificial intelligence to | | | , , |
| Ming- | analyze 24-hour esophageal pH-impedance | | 2022/1/1~ | Hualien Tzu |
| Wen | monitoring: Technological efficacy and clinical | Principal Investigator | $2022/1/1$ $\approx$ $2022/12/31$ | Chi Hospital |
| | applications in the diagnosis of gastroesophageal reflux disease (GERD). | | | <b></b> |
| Weng | The therapeutic effects of concentrated Jingsu | C D: : 1 | 2022/01/01 | Tzu Chi |
| Ming- | herbal drink on physical and psychological | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Medical |
| Wen | symptoms of long COVID—gut-brain axis | mvestigatoi | 2023/12/31 | Foundation |

| | Version Date: (Version 8, 11/19/2024) | | _ | |
|---|---|---|---|---|
| | dysregulation: A randomized double-blind clinical trial. | | | |
| Weng<br>Ming-<br>Wen | Exploring the interplay between belching, psychological symptoms, and esophageal acid reflux: Clinical applications for optimizing the treatment of gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | Exploring the pathophysiological role and interplay of esophageal hypersensitivity, psychological distress, and functional gastrointestinal disorders in patients with esophageal symptoms. | Co-Principal | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | Analyzing the pharyngeal swallowing physiology in patients with ineffective esophageal motility using high-resolution pharyngeal function testing. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | Exploring the relationship between esophageal capsaicin sensitivity, motility sensation, and physiological features of reflux: Clinical impacts and treatment guidelines for esophageal dysfunction and gastroesophageal reflux disease (GERD). | Co-Principal<br>Investigator | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Weng<br>Ming-<br>Wen | The application of high-resolution impedance pharyngeal function testing and the Sydney Swallowing Questionnaire in the assessment of oropharyngeal swallowing difficulties and voice disorders. | Co-Principal | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | The application of artificial intelligence in high-<br>resolution esophageal function testing: A study<br>using an unsupervised deep learning-based<br>algorithm model. | | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | Exploring the clinical characteristics and the impact of gut microbiota in patients with metabolic-associated fatty liver disease under dietary and exercise regulation. | Co-Principal | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | The therapeutic effects of Jing Si Herbal Drink on<br>the psychosomatic symptoms of functional<br>dyspepsia: A randomized double-blind clinical<br>trial. | | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Foundation |
| Weng<br>Ming-<br>Wen | The use of proximal esophageal nocturnal average baseline mucosal impedance values to improve the diagnosis of laryngopharyngeal reflux disease and establish indications for proton pump inhibitors. | Principal Investigator | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Weng<br>Ming-<br>Wen | The exploration of the pathophysiological impact of esophageal contraction, mucosal integrity, and acid sensitivity on gastroesophageal reflux disease, along with therapeutic strategies based on these factors. | Co-Principal<br>Investigator | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Weng<br>Ming-<br>Wen | Exploring the role of esophageal microbiota in gastroesophageal reflux disease through novel impedance parameters, clinical classification, and hypersensitivity. | Co-Principal | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Weng<br>Ming-<br>Wen | Exploring the relationship and pathophysiological mechanisms between esophageal acid sensitivity, secondary esophageal contraction, and subtypes of gastroesophageal reflux disease. | Co-Principal | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |

| | Version Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| Weng<br>Ming- | Exploring the clinical application of high-<br>resolution impedance pharyngoesophageal | Co-Principal | 2021/1/1~ | Hualien Tzu |
| Wen | function testing in the assessment of pharyngeal dysphagia and drug responses. | Investigator | 2021/12/31 | Chi Hospital |
| Yi Zhi-<br>Xun | The efficacy of Jing's Herbal Decoction Concentrate in treating long COVID symptoms—gut-brain axis dysfunction and associated physical and mental symptoms: A randomized double-blind clinical trial. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Foundation |
| Yi Zhi-<br>Xun | Exploring the interaction between belching, physical and mental symptoms, and esophageal acid reflux: Clinical applications for optimizing gastroesophageal reflux disease treatment. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Exploring the pathophysiological mechanisms and interactions of esophageal hypersensitivity, psychological distress, and functional gastrointestinal disorders in patients with esophageal symptoms. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Exploring the efficacy and physiological changes of anti-reflux mucosal ablation therapy in proton pump inhibitor-dependent gastroesophageal reflux disease. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Analyzing the pharyngeal swallowing physiology and dynamics in patients with ineffective esophageal motility using high-resolution pharyngoesophageal function testing. | Co-Principal<br>Investigator | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Exploring the relationship between esophageal capsaicin sensitivity, motility sensory function, and the reflux characteristics of physical and psychological physiology: Clinical impact and treatment guidelines for esophageal dysfunction and gastroesophageal reflux disease. | Co-Principal<br>Investigator | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology<br>(MOST) |
| Yi Zhi-<br>Xun | Exploring the pathophysiological mechanisms of gastroesophageal reflux disease through esophageal clearance ability, mucosal integrity, and psychological characteristics, and establishing the basis for precise diagnosis and treatment. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Exploring the impact of opioid analgesics on the pathophysiological mechanisms of esophageal contraction and reflux characteristics, and their clinical applications. | Co-Principal<br>Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | The application of high-resolution impedance pharyngoesophageal function testing and the Sydney Swallow Questionnaire in oropharyngeal dysphagia and voice disorders. | Co-Principal | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | The Application of Artificial Intelligence in High-Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. | Investigator | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi Zhi-<br>Xun | Artificial Intelligence Analysis of 24-Hour Esophageal pH Impedance Testing Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. | Co-Principal | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |

| | ersion Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| Yi Zhi- | Exploring the Impact of Diet and Exercise | | | |
| Xun | Regulation on Clinical Features and Gut | Co-Principal 2022/1/1~ | | Hualien Tzu |
| | Microbiota in Patients with Metabolism-Related | Investigator | 2022/12/31 | Chi Hospital |
| | Fatty Liver Disease. | 5 | | 1 |
| Yi Zhi- | The Therapeutic Effect of Jinseng Herbal Drink on | | | T ~1. |
| Xun | Psychosomatic Symptoms in Functional | Co-Principal | 2022/1/1~ | Tzu Chi |
| 2 2 2011 | Dyspepsia: A Randomized Double-Blind Clinical | Investigator | 2022/17/1 | Medical |
| | Trial. | mvestigator | 2022/12/J1 | Foundation |
| Yi Zhi- | | | | |
| | Exploring the Interrelationship and Pathogenic | | 2021/1/1 | II11 |
| Xun | Mechanisms Between Esophageal Acid Sensitivity, | Principal Investigator | 2021/1/1~ | Hualien Tzu |
| | Esophageal Secondary Contractions, and Subtypes | 1 10020 | 2021/12/31 | Chi Hospital |
| | of Gastroesophageal Reflux Disease. | | | |
| Yi Zhi- | Exploring the Role of Esophageal Microbiota in | | | |
| Xun | Gastroesophageal Reflux Disease: Its Impact on | Co-Principal | 2021/1/1~ | Hualien Tzu |
| | Novel Impedance Parameters, Clinical | Investigator | 2021/12/31 | Chi Hospital |
| | Classification, and Hypersensitivity. | Č | | • |
| Yi Zhi- | Clinical Application of High-Resolution | | | |
| Xun | Impedance Pharyngeal Function Testing in the | Co-Principal | 2021/1/1~ | Hualien Tzu |
| 2 2 2011 | Assessment of Pharyngeal Dysphagia and Drug | Investigator | 2021/17/1 | Chi Hospital |
| | Response. | mvestigator | 2021/12/J1 | om Hospital |
| Yi Zhi- | 1 | | | Ministerraf |
| | Exploring the Pathophysiological Impact of | Ca Duin i 1 | 2020/0/1 | Ministry of |
| Xun | Esophageal Contractions, Mucosal Integrity, and | Co-Principal | 2020/8/1~ | Science and |
| | Acid Sensitivity on Gastroesophageal Reflux | Investigator | 2023/07/31 | Technology |
| | Disease and the Basis for Therapeutic Strategies. | | | (MOST) |
| Liu Zuo- | Exploring the Impact of Diet and Exercise | | | |
| Cai | Regulation on Clinical Features and Gut | Principal Investigator | 2022/1/1~ | Hualien Tzu |
| | Microbiota in Patients with Metabolism-Related | i imcipai mvestigatoi | 2022/12/31 | Chi Hospital |
| | Fatty Liver Disease. | | | |
| Liu Zuo- | The Therapeutic Effect of Jinseng Herbal Extract | | | |
| Cai | on Long COVID Symptoms: Psychosomatic | O D : 1 | 2022/01/01 | Tzu Chi |
| | Symptoms Related to Gut-Brain Axis | Co-Principal | 2023/01/01~ | Medical |
| | Dysregulation – A Randomized Double-Blind | Investigator | 2023/12/31 | Foundation |
| | Clinical Trial. | | | 1 Candation |
| Liu Zuo- | Exploring the Interrelationship Between Belching, | | | |
| | | Co. Duin ain -1 | 2022/01/01 | Huolian T- |
| Cai | Psychosomatic Symptoms, and Esophageal Acid | <u>=</u> | 2023/01/01~ | Hualien Tzu |
| | Reflux: Clinical Applications for Optimizing | Investigator | 2023/12/31 | Chi Hospital |
| | Gastroesophageal Reflux Disease Treatment. | | | |
| Liu Zuo- | Exploring the Pathophysiological Mechanisms and | | | |
| Cai | Interrelationship Between Esophageal | Co-Principal | 2023/01/01~ | Hualien Tzu |
| | Hypersensitivity, Psychological Distress, and | - | 2023/01/01~ | Chi Hospital |
| | Functional Gastrointestinal Disorders in Patients | Investigator | 2023/12/31 | Ciii nospital |
| | with Esophageal Symptoms. | | | |
| Liu Zuo- | Analyzing the Pharyngeal Physiology and | | | |
| Cai | Dynamics of Swallowing in Esophageal Ineffective | Co-Principal | 2023/01/01~ | Hualien Tzu |
| Cui | Peristalsis Patients Using High-Resolution | Investigator | 2023/01/01~ | Chi Hospital |
| | | mvestigator | 2023/12/31 | em Hospital |
| Lin 7: | Pharyngeal Function Testing. | | | |
| Liu Zuo- | Exploring the Efficacy and Physiological Changes | | 2022/01/01 | II 1' T |
| Cai | of Anti-Reflux Mucosal Ablation in Proton Pump | Co-Principal | 2023/01/01~ | Hualien Tzu |
| | Inhibitor-Dependent Gastroesophageal Reflux | Investigator | 2023/12/31 | Chi Hospital |
| | Disease. | | | |
| Liu Zuo- | Exploring Esophageal Capsaicin Sensitivity, | | | Ministry of |
| Cai | Peristaltic Sensory Function, and | Co-Principal | 2023/8/1~ | Science and |
| | Psychophysiological Reflux Characteristics: | Investigator | 2026/07/31 | Technology |
| | Clinical Impact and Treatment Guidelines for | C | | (MOST) |
| | TT Sales Treatment Galacinies 101 | | | () |

| v | ersion Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|
| | Esophageal Dysfunction and Gastroesophageal | | | |
| | Reflux Disease. | | | |
| Liu Zuo- | Exploring the Pathophysiological Mechanisms of | | | |
| Cai | Gastroesophageal Reflux Disease Through | | | |
| Cai | Esophageal Reflux Clearance Ability, Mucosal | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | 1 1 0 | Investigator | 2022/12/31 | Chi Hospital |
| | Integrity, and Psychosocial Traits: Establishing the | C | | • |
| | Basis for Precise Diagnosis and Treatment. | | | |
| Liu Zuo- | Exploring the Impact of Opioid Analgesics on | | | |
| Cai | Esophageal Contraction and Reflux | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | Characteristics: Pathophysiological Mechanisms | Investigator | 2022/12/31 | Chi Hospital |
| | and Clinical Applications. | C | | 1 |
| Liu Zuo- | The Application of High-Resolution Impedance | | | |
| Cai | Pharyngeal Function Testing and the Sydney | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Cai | Swallowing Questionnaire in Oropharyngeal | Investigator | 2022/17/1 | Chi Hospital |
| | | mvestigator | 2022/12/31 | Cili Hospitai |
| 1 . 7 | Dysphagia and Voice Disorders. | | | |
| Liu Zuo- | Artificial Intelligence Analysis of 24-Hour | | | |
| Cai | Esophageal pH-Impedance Monitoring Using | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | Supervised Learning: Technical Performance and | Investigator | 2022/12/31 | Chi Hospital |
| | Clinical Applications in the Diagnosis of | mvestigator | 2022/12/31 | Cm Hospital |
| | Gastroesophageal Reflux Disease. | | | |
| Liu Zuo- | The Application of Artificial Intelligence in High- | | | |
| Cai | Resolution Esophageal Function Testing: A Study | Co-Principal | 2022/1/1~ | Hualien Tzu |
| | on Unsupervised Computational Models Based on | Investigator | 2022/12/31 | Chi Hospital |
| | Deep Learning. | in vestigater | 2022/12/01 | em Hospital |
| Liu Zuo- | The Therapeutic Effect of Jinseng Herbal Drink on | | | |
| Cai | | | 2022/1/1~ | Tzu Chi |
| Cai | J 1 | Co-Principal | | Medical |
| | Dyspepsia: A Randomized Double-Blind Clinical Trial. | Investigator | 2022/12/31 | Foundation |
| Liu Zuo- | Exploring the Role of Esophageal Microbiota in | | | |
| | | | 2021/1/1~ | Hualien Tzu |
| Cai | Gastroesophageal Reflux Disease: Its Impact on | Co-Principal | | |
| | Novel Impedance Parameters, Clinical | Investigator | 2021/12/31 | Chi Hospital |
| | Classification, and Hypersensitivity. | | | |
| Liu Zuo- | Exploring the Interrelationship and Pathogenic | | | |
| Cai | Mechanisms Between Esophageal Acid Sensitivity, | Co-Principal | 2021/1/1~ | Hualien Tzu |
| | Esophageal Secondary Contractions, and Subtypes | Investigator | 2021/12/31 | Chi Hospital |
| | of Gastroesophageal Reflux Disease. | | | |
| Liu Zuo- | Clinical Application of High-Resolution | | | |
| Cai | Impedance Pharyngeal Function Testing in the | Co-Principal | 2021/1/1~ | Hualien Tzu |
| | Assessment of Pharyngeal Dysphagia and Drug | Investigator | 2021/12/31 | Chi Hospital |
| | Response. | in vestigator | 2021/12/31 | em Hospital |
| Liu Zuo- | Exploring the Pathophysiological Impact of | | | Ministry of |
| | | Co Duin oin al | 2020/8/1~ | Science and |
| Cai | Esophageal Contractions, Mucosal Integrity, and | Co-Principal | | |
| | Acid Sensitivity on Gastroesophageal Reflux | Investigator | 2023/07/31 | Technology |
| | Disease and the Basis for Therapeutic Strategies. | | | (MOST) |
| Hong | Analyzing the Pharyngeal Physiology and | | | |
| Rui- | Dynamics of Swallowing in Esophageal Ineffective | Principal Investigator | 2023/01/01~ | Hualien Tzu |
| Sheng | Peristalsis Patients Using High-Resolution | i imorpai investigatoi | 2023/12/31 | Chi Hospital |
| | Pharyngeal Function Testing. | | | - |
| Hong | The Application of High-Resolution Impedance | | | |
| Rui- | Pharyngeal Function Testing and the Sydney | | 2022/1/1~ | Hualien Tzu |
| Sheng | Swallowing Questionnaire in Oropharyngeal | Principal Investigator | 2022/12/31 | Chi Hospital |
| Silving | Dysphagia and Voice Disorders. | | 2022/12/31 | om mospitui |
| | Dyspilagia aliu voice Districts. | | | |

| | Version Date: (Version 8, 11/19/2024) | | 1 | |
|---|---|---|---|---|
| Hong | The Therapeutic Effect of Jinseng Herbal Extract | | | |
| Rui- | on Long COVID Symptoms: Psychosomatic | Ca Principal | 2022/01/01 | Tzu Chi |
| Sheng | Symptoms Related to Gut-Brain Axis | Co-Principal | 2023/01/01~ | Medical |
| | Dysregulation – A Randomized Double-Blind | Investigator | 2023/12/31 | Foundation |
| | Clinical Trial. | | | 1 0 00000000000000000000000000000000000 |
| Hong | Exploring the Interrelationship Between Belching, | | | |
| Rui- | 1 | Co Principal | 2022/01/01 | Hualien Tzu |
| | Psychosomatic Symptoms, and Esophageal Acid | - | 2023/01/01~ | |
| Sheng | Reflux: Clinical Applications for Optimizing | Investigator | 2023/12/31 | Chi Hospital |
| | Gastroesophageal Reflux Disease Treatment. | | | |
| Hong | Exploring the Pathophysiological Mechanisms and | | | |
| Rui- | Interrelationship Between Esophageal | Co-Principal | 2023/01/01~ | Hualien Tzu |
| Sheng | Hypersensitivity, Psychological Distress, and | * | 2023/01/01~ | |
| | Functional Gastrointestinal Disorders in Patients | Investigator | 2023/12/31 | Chi Hospital |
| | with Esophageal Symptoms. | | | |
| Hong | Exploring the Efficacy and Physiological Changes | | | |
| Rui- | of Anti-Reflux Mucosal Ablation in Proton Pump | Co-Principal | 2023/01/01~ | Hualien Tzu |
| Sheng | Inhibitor-Dependent Gastroesophageal Reflux | Investigator | 2023/01/01 | Chi Hospital |
| Sheng | 1 | mvestigator | 2023/12/31 | Cili Hospital |
| T T | Disease. | | | |
| Hong | Exploring Esophageal Capsaicin Sensitivity, | | | 3.51 |
| Rui- | Peristaltic Sensory Function, and | | | Ministry of |
| Sheng | Psychophysiological Reflux Characteristics: | Co-Principal | 2023/8/1~ | Science and |
| | Clinical Impact and Treatment Guidelines for | Investigator | 2026/07/31 | Technology |
| | Esophageal Dysfunction and Gastroesophageal | _ | | (MOST) |
| | Reflux Disease. | | | , |
| Hong | Exploring the Pathophysiological Mechanisms of | | | |
| Rui- | Gastroesophageal Reflux Disease Through | | | |
| Sheng | Esophageal Reflux Clearance Ability, Mucosal | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Sheng | | Investigator | 2022/12/31 | Chi Hospital |
| | Integrity, and Psychosocial Traits: Establishing the | | | - |
| ** | Basis for Precision Diagnosis and Treatment. | | | |
| Hong | Exploring the Impact of Opioid Analgesics on | | | |
| Rui- | Esophageal Contraction and Reflux | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Sheng | Characteristics: Pathophysiological Mechanisms | Investigator | 2022/12/31 | Chi Hospital |
| | and Clinical Applications. | | | |
| Hong | Artificial Intelligence Analysis of 24-Hour | | | |
| Rui- | Esophageal pH-Impedance Monitoring Using | | 0000/1/4 | ** 11 |
| Sheng | Supervised Learning: Technical Performance and | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Sheng | Clinical Applications in the Diagnosis of | Investigator | 2022/12/31 | Chi Hospital |
| | Gastroesophageal Reflux Disease. | | | |
| Hama | The Application of Artificial Intelligence in High- | | | |
| Hong | | C. D. in a in a 1 | 2022/1/1 | П1: Т |
| Rui- | Resolution Esophageal Function Testing: A Study | | 2022/1/1~ | Hualien Tzu |
| Sheng | on Unsupervised Computational Models Based on | Investigator | 2022/12/31 | Chi Hospital |
| | Deep Learning. | | | |
| Hong | Exploring the Impact of Diet and Exercise | | | |
| Rui- | Regulation on Clinical Features and Gut | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Sheng | Microbiota in Patients with Metabolism-Related | Investigator | 2022/12/31 | Chi Hospital |
| | Fatty Liver Disease. | | | • |
| Hong | The Therapeutic Effect of Jinseng Herbal Drink on | | | T. ~: |
| Rui- | Psychosomatic Symptoms in Functional | Co-Principal | 2022/1/1~ | Tzu Chi |
| Sheng | Dyspepsia: A Randomized Double-Blind Clinical | | 2022/17/17 | Medical |
| Shelig | Trial. | mvestigatoi | 4044/14/31 | Foundation |
| II | | | | |
| Hong | Clinical Application of High-Resolution | | 2021/1/1 | II 1' T |
| Rui- | Impedance Pharyngeal Function Testing in the | Principal Investigator | 2021/1/1~ | Hualien Tzu |
| Sheng | Assessment of Oropharyngeal Dysphagia and Drug | 1 : 557551 | 2021/12/31 | Chi Hospital |
| | Response. | | | |

| Rui- Sheng Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Hong Exploring the Interrelationship and Pathogenic Rui- Sheng Exploring the Interrelationship and Pathogenic Pat | v | Yersion Date: (Version 8, 11/19/2024) | | | |
|---|---|---|---|---|---|
| Sheng Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. | Hong | Exploring the Role of Esophageal Microbiota in | | | |
| Classification, and Hypersensitivity. Rui Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Hong Rui-Sheng Exploring the Pathophysiological Impact of Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. Liang Bhu-Wei Exploring the Pathophysiological Impact of Esophageal Computational Models Based on Deep Learning. Artificial Intelligence Analysis of 24-Hour Supervised Computational Models Based on Deep Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Triatis: Establishing the Basis for Precision Diagnosis and Treatment. Exploring the Impact of Opioid Analgesics on Schageal phenoment of Co-Principal Investigator (Co-Principal In | Rui- | Gastroesophageal Reflux Disease: Its Impact on | Co-Principal | 2021/1/1~ | Hualien Tzu |
| Classification, and Hypersensitivity. Rui Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Hong Rui-Sheng Exploring the Pathophysiological Impact of Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. Liang Bhu-Wei Exploring the Pathophysiological Impact of Esophageal Computational Models Based on Deep Learning. Artificial Intelligence Analysis of 24-Hour Supervised Computational Models Based on Deep Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Triatis: Establishing the Basis for Precision Diagnosis and Treatment. Exploring the Impact of Opioid Analgesics on Schageal phenoment of Co-Principal Investigator (Co-Principal In | Sheng | Novel Impedance Parameters, Clinical | - | 2021/12/31 | Chi Hospital |
| Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Co-Principal Investigator 2021/12/31 Chi Hospital Disease and the Basis for Therapeutic Strategies. Co-Principal Investigator 2023/07/31 Technology (MOST) Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. The Application of Artificial Intelligence in High-Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. The Applications of Artificial Intelligence Analysis of 24-Hour Esophageal pH-Impedance Monitoring Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Co-Principal Investigator 2022/12/31 Chi Hospital Investigator 2022/12/31 Co-Principal Investigator 2022/12/31 Chi Hospital Co-Principal Investigator 2022/12/31 Co-Principal Investigator 2022/12/31 Chi Hospital Co-Principal Investigator 2021/12/31 Chi Hospital Co-Principal Investigator 2021/12/31 Chi Hosp | | Classification, and Hypersensitivity. | C | | 1 |
| Mechanisms Between Isophageal Acid Sensitivity. Co-Principal 2021/11- Univestigator of Gastroesophageal Reflux Disease. Co-Principal 2021/12/31 Chi Hospital | Hong | | | | |
| Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Co-Principal Disease and the Basis for Therapeutic Strategies. Co-Principal Disease and the Basis for Therapeutic Strategies. Co-Principal Disease and the Basis for Therapeutic Strategies. Co-Principal Disease and the Basis for Therapeutic Strategies. Principal Investigator Co-Principal Disease and the Basis for Therapeutic Strategies. Principal Disease and the Basis for Therapeutic Strategies. Principal Investigator Co-Principal Disease Dise | Rui- | | Co-Principal | 2021/1/1~ | Hualien Tzu |
| of Gastroesophageal Reflux Disease. Hong Exploring the Pathophysiological Impact of Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. Liang Shu-Wei Contraction of Artificial Intelligence in High-Resolution Esophageal Function Testing: A Study on Deep Learning. Artificial Intelligence Analysis of 24-Hour Esophageal Reflux Disease. Liang Shu-Wei Contraction in the Diagnosis of Gastroesophageal Reflux Disease. Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Esophageal Reflux Disease. Liang Exploring the Impact of Opioid Analgesics on Foophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Exploring the Impact of Opioid Analgesics on Foophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Exploring the Impact of Diet and Exercise Regulation on Clinical Evaluation of Clinical Applications. Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Role of Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Louisidator Co-Principal Louisi | Sheng | _ = = | - | 2021/12/31 | Chi Hospital |
| Exploring the Pathophysiological Impact of Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. | 8 | 1 0 1 | 8 | | 1 |
| Esophageal Contractions, Mucosal Integrity, and Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. Liang Shu-Wei Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Shu-Wei Esophageal PH-Impedance Monitoring Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease. Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Fatty Liver Disease. Liang Shu-Wei Exploring the Impact of Diet and Exercise Fatty Liver Disease. Liang Shu-Wei Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Role of Esophageal Reflux Disease. Clinical Appli | Hong | ž - Ū | | | Ministry of |
| Sheng Acid Sensitivity on Gastroesophageal Reflux Disease and the Basis for Therapeutic Strategies. Liang Shu-Wei Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. Liang Shu-Wei Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Shu-Wei Regulation on Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Exploring the Role of Esophageal Microbiota in Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Resulting Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Responsable Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Reflux Disease: Liang Clinical Applications of High-Resolution Impedance Pharyngeal Psysphagia and Drug Investigator 2021/11/2 Investigator 2021/11/2 Investigator 2021/11/2 Investigator 2021/11/2 Chi Hospital Chi Hospital Investigator 2021/11/2 Chi Hospital Chi-Co-Principal Investigator 2021/12/3 Chi Hospital Chi-Co-Principal Investigator 2021/11/2 Chi Hospital Chi-Co-Principal Investigator 2021/11/2 Chi Hospital Chi-Co-Principal Investigator 2021/11/2 Chi Hospital Chi-Co-Principal 2021/11/2 Chi Hospital Chi-Co-Principal 2021/11/2 Chi Hospital C | Rui- | | Co-Principal | 2020/8/1~ | |
| Disease and the Basis for Therapeutic Strategies. Liang Shu-Wei Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. Liang Shu-Wei Esophageal pH-Impedance Monitoring Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Shu-Wei Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Exploring the Impact of Opioid Analgesics on Esqualition on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Muchanisms Between Esophageal Reflux Disease. Classification, and Hypersensitivity. Ecophageal Contractions, and Subtypes of Gastroesophageal Reflux Disease. Clinical Application of High-Resolution Impedance Pharyngeal Purction Testing in the Pathopatha Pa | | | <u>=</u> | | |
| The Application of Artificial Intelligence in High- Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. Liang | | | | | 0. |
| Shu-Wei Resolution Esophageal Function Testing: A Study on Unsupervised Computational Models Based on Deep Learning. Liang Artificial Intelligence Analysis of 24-Hour Esophageal pH-Impedance Monitoring Using Shu-Wei Esophageal pH-Impedance Monitoring Using Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Disease. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Disease. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Function Testing in the Machanisms Tental Tru Chi Hualien Tzu Chi Hospital Tru Chi Hualien Tzu Chi Hualien Tzu Chi Hospital Tru Chi Hualien Tz | Liano | | | | (1.1021) |
| on Unsupervised Computational Models Based on Deep Learning. Liang Shu-Wei Esophageal PH-Impedance Monitoring Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Disease Through Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Shu-Wei Esophageal Reflux Clearaction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Gastroesophageal Reflux Disease Through Exploring the Impact of Diet and Exercise Fatty Liver Disease. Liang Shu-Wei Gastroesophageal Reflux Classification, and Hypersensitivity. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/1/1- Hualien Tzu Chi Hospital Co-Principal 2021/1/1- Hualien Tzu Chi Hospital Co-Princip | _ | •• | | 2022/1/1~ | Hualien Tzu |
| Deep Learning. | Sila Wei | 1 0 | Principal Investigator | | |
| Co-Principal Co-P | | | | 2022/12/31 | Cili Hospital |
| Shu-Wei Esophageal pH-Impedance Monitoring Using Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Shu-Wei Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Shu-Wei Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Postenses and Exploring the Role of Esophageal Microbiota in Postenses and Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Postenses and Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Postenses and Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Postenses and Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Postenses and Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Shu-Wei Role of Esophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Esophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Col-Principal 2021/11/~ Hualien Tzu Chi Hospital Chi Hospital Col-Principal 2021/11/~ Hualien Tzu Chi Hospital Ch | Liona | | | | |
| Supervised Learning: Technical Performance and Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Shu-Wei Esophageal Contraction and Reflux Chiracteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Shu-Wei Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interventions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Punction Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2022/11/2/31 Chi Hospital Co-Principal 2022/11/2/31 Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Chi Hospital Co-Principal 2021/11/2/31 Chi Hospital Chi Hospita | | Esophageal pH Impedance Manitoring Using | | | |
| Clinical Applications in the Diagnosis of Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Role of High-Resolution of High-Resolution Impedance Pharyngeal Psyphagia and Drug Log21/12/31 Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Psu-Wei Psychosomatic Symptoms in Functional Dyspesia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Chi | Silu- WCI | | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Gastroesophageal Reflux Disease. Liang Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Gastroesophageal Reflux Disease: Its Impact on Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hualien Tzu Chi Hospital | | = | Investigator | 2022/12/31 | Chi Hospital |
| Exploring the Pathophysiological Mechanisms of Gastroesophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Shu-Wei Exploring the Impact of Diet and Exercise Fatty Liver Disease. Liang Exploring the Impact of Diet and Exercise Fatty Liver Disease. Liang Exploring the Role of Esophageal Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Co-Principal Investigator 2022/11/~ Chi Hospital Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Its Impact on Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Interpretation Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Hualien Tzu Chi Hospital Co-Principal Co- | | 1 11 | | | |
| Shu-Wei Gastroesophageal Reflux Disease Through Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Shu-Wei Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Shu-Wei Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Off Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Chimage Characteristics Pathophysiological Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Its Impact on Co-Principal Investigator Pathogenic Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease: Interpretationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Reflux Disease: Interpretation of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Chi Hospital Chi Hospital Chi Hospital Chi Hospital Chi Hospital Ch | T iama | | | | |
| Esophageal Reflux Clearance Ability, Mucosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Shu-Wei Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Shu-Wei Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Gastroesophageal Reflux Disease. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital 2021/1/1/2 C | | | | | |
| Investigator Sophageal Reflux Clearance Ability, Micosal Integrity, and Psychosocial Traits: Establishing the Basis for Precision Diagnosis and Treatment. | Snu-wei | | Co-Principal | 2022/1/1~ | Hualien Tzu |
| Basis for Precision Diagnosis and Treatment. Liang Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Shu-Wei Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Dyschosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Punction Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Chi Hospital Investigator 2021/12/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Chineal Application of High-Resolution Impedance Pharyngeal Punction Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Chi Hospital | | | <u>=</u> | 2022/12/31 | Chi Hospital |
| Exploring the Impact of Opioid Analgesics on Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2022/1/1~ Hualien Tzu Chi Medical Foundation Co-Principal 2021/1/1~ Hualien Tzu Chi Medical Foundation Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Chi Hospital Co-Principal 2021/1/1/2 Chi Hospital Co-Principal 2021/1/1/2 Chi Hospital Co-Principal 2021/1/1/2 Chi Hospital | | | C | | 1 |
| Shu-Wei Esophageal Contraction and Reflux Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Chi Hospital Co-Principal 2021/11/~ Chi Hospital Chi Hospital Chi Hospital Chi Hospital Co-Principal Investigator 2021/12/31 Chi Hospital Ch | т • | | | | |
| Characteristics: Pathophysiological Mechanisms and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Liang Clinical Application Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Liang Clinical Application Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Liang Clinical Application Oropharyngeal Dysphagia and Drug Investigator Liang Clinical Ap | | = = = | G D: : 1 | 2022/4/4 | TT 1' T |
| and Clinical Applications. Liang Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Impedance Parameters Clinical Classification, and Hypersensitivity. Liang Exploring the Impedance Parameters Clinical Classification of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Ch | Shu-Wei | 1 6 | * | | |
| Exploring the Impact of Diet and Exercise Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Shu-Wei Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Is Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2022/1/1~ Tzu Chi Medical Foundation Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital | | 1 | Investigator | 2022/12/31 | Chi Hospital |
| Shu-Wei Regulation on Clinical Features and Gut Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Dyspensia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Cassification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Co-Principal 2022/11/~ Medical Tzu Chi Medical Foundation Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Chi Hospital Co-Principal 2021/11/~ Chi Hospital Co-Principal 2021/11/~ Chi Hospital Co-Principal 2021/11/~ Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Chi Hospital | | | | | |
| Microbiota in Patients with Metabolism-Related Fatty Liver Disease. Liang Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Microbiota in Patients with Metabolism-Related Investigator Co-Principal 2022/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital | | | 1 1 1 | | 4. – |
| Fatty Liver Disease. Liang The Therapeutic Effect of Jinseng Herbal Drink on Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11~ Hualien Tzu Co-Principal 2021/11/2 Hualien Tzu Co-Principal 2021/11/31 Chi Hospital Co-Principal 2021/12/31 Chi Hospital Co-Principal 2021/11/31 Chi Hospital | Shu-Wei | | | | |
| Liang Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Chi Hospital | | | Investigator | 2022/12/31 | Chi Hospital |
| Shu-Wei Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11~ Hualien Tzu Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital Co-Principal 2021/12/31 Chi Hospital Chi Hospital | | | | | |
| Psychosomatic Symptoms in Functional Dyspepsia: A Randomized Double-Blind Clinical Trial. | _ | 1 | | | Tzu Chi |
| Dyspepsia: A Randomized Double-Blind Clinical Trial. Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Divestigator 2021/1/1~ Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Hualien Tzu Chi Hospital Co-Principal 2021/11/2 Chi Hospital Co-Principal 2021/11/2 Chi Hospital Chi Hospital | Shu-Wei | ] ] ] | <u>=</u> | | |
| Liang Exploring the Role of Esophageal Microbiota in Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/1 Chi Hospital | | 7 = = | Investigator | 2022/12/31 | |
| Shu-Wei Gastroesophageal Reflux Disease: Its Impact on Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Chi Hospital | | | | | Toundation |
| Novel Impedance Parameters, Clinical Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11/1~ Hualien Tzu 2021/11/1~ Hualien Tzu 2021/11/1 Chi Hospital Co-Principal 2021/11/1 Chi Hospital Co-Principal 2021/11/1 Chi Hospital Co-Principal 2021/11/1 Chi Hospital Chi Hospital | | | | | |
| Classification, and Hypersensitivity. Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Hualien Tzu Investigator 2021/12/31 Chi Hospital | Shu-Wei | 1 1 | <u>=</u> | | |
| Liang Exploring the Interrelationship and Pathogenic Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Chi Hospital | | Novel Impedance Parameters, Clinical | Investigator | 2021/12/31 | Chi Hospital |
| Shu-Wei Mechanisms Between Esophageal Acid Sensitivity, Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Co-Principal 2021/11/~ 2021/12/31 Chi Hospital Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Hualien Tzu Co-Principal 2021/11/~ Chi Hospital | | | | | |
| Esophageal Secondary Contractions, and Subtypes of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital Co-Principal 2021/11/2 Hualien Tzu 2021/12/31 Chi Hospital | Liang | = = = | | | |
| of Gastroesophageal Reflux Disease. Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator October 1 | Shu-Wei | 1 2 | Co-Principal | 2021/1/1~ | Hualien Tzu |
| Liang Clinical Application of High-Resolution Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator Co-Principal 2021/1/1~ Hualien Tzu Investigator 2021/12/31 Chi Hospital | | | Investigator | 2021/12/31 | Chi Hospital |
| Shu-Wei Impedance Pharyngeal Function Testing in the Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/11/2 Hualien Tzu 2021/12/31 Chi Hospital | | of Gastroesophageal Reflux Disease. | | | |
| Assessment of Oropharyngeal Dysphagia and Drug Investigator 2021/12/31 Chi Hospital | Liang | Clinical Application of High-Resolution | | | |
| | Shu-Wei | Impedance Pharyngeal Function Testing in the | Co-Principal | 2021/1/1~ | Hualien Tzu |
| Response. | | Assessment of Oropharyngeal Dysphagia and Drug | Investigator | 2021/12/31 | Chi Hospital |
| | | Response. | | | |

## 5. Research Related to Costs

| | Project Name | Description | Unit Price (NTW) | Quantity | Total Price (NTW) | Remarks |
|---|---|---|---|---|---|---|
| | 1.Research Personnel Costs (For related insurance premiums, please consult the Human Resources Department) | <ul> <li>(1) Full-time Personnel (for individual project applications only):</li> <li>Work remuneration (including year-end bonus reserve)</li> <li>Employer contribution to labor and health insurance</li> <li>Employer contribution to labor pension (6% of insured salary)</li> </ul> | | | | |
| 1. Operational Expenses | | (2) Part-time Personnel (must be enrolled students): • Work remuneration □ Undergraduate student □ Master's student □ Other: • Employer contribution to labor and health insurance • Employer contribution to labor pension (6% of insured salary) (3) Temporary Workers: • Work remuneration • Employer contribution to labor and health insurance • Employer contribution to labor pension (6% of insured salary) (4) Professional Assistance Fees | | 40 | 480,000 | |
| | 2 Amires al | rees | | Subtotal: | 480,000 | |
| | 2.Animal Experimentation Fees | | | Subtotal: | | |
| | 3.Consumables,<br>Equipment,<br>Books, and<br>Miscellaneous<br>Expenses | Participant Stipends Miscellaneous: Postage and Telecommunications, Printing Costs, Copy Paper, Copying | 500<br>1,000<br>15,000 | 40 | Í | |

| Version Date : (Version 8 | , 11/19/2024) | | | |
|---|---|---|---|---|
| | Fees, Binding Fees, Stationery | | | |
| | Costs, Poster Production Fees, | | | |
| | Computer Data Statistics Fees, | | | |
| | Computer Data Analysis Fees, | | | |
| | Paper Submission Fees, Paper | | | |
| | Publication Fees, Sectioning, | | | |
| | Embedding, and Staining | | | |
| | Immunology Costs. | | | |
| | | Subt | total: | 160,000 |
| 2. Research | | | | |
| <b>Equipment Costs</b> | | | | |
| (According to | | | | |
| regulations, books, | | | | |
| computers, and | | | | |
| peripheral equipment | | Subt | total: | 0 |
| are not included in the | | | | |
| subsidy. Medium and | | | | |
| large instruments will | | | | |
| be applied for | | | | |
| collectively by the | | | | |
| research department, | | | | |
| based on necessity, | | | | |
| for shared use.) | | | | |
| | Total | | | 640,000 |

### 6. Project Abstract

( Please provide a summary of the key points of this project within 500 words, and create customized keywords based on the nature of the project.)

Gastroesophageal reflux disease (GERD) poses a challenging medical condition to manage, with up to 40% of patients showing refractory to standard medical intervention, which usually begins with a proton pump inhibitor (PPI). Among these cases, esophageal disorders of gut-brain interaction (DGBI), such as reflux hypersensitivity and functional heartburn, or GERD patients with concurrent occurrences of these conditions, constitute more than 90% of the patients who did not respond to twice-daily PPI treatment. Esophageal visceral hypersensitivity and hypervigilance are the two pathways that drive esophageal DGBI and symptoms. The Rome IV esophageal disorders, encompassing functional chest pain, functional heartburn, globus, functional dysphagia, and reflux hypersensitivity, are defined by present with symptoms originating from the esophagus without detectable evidence of structural, inflammatory, or motor disorders. Diagnosing esophageal DGBI necessitates testing involving endoscopy, pH-impedance monitoring, and high-resolution manometry. Neuromodulators form the basis of the pharmacological strategy for managing various esophageal DGBI and symptoms, modulating both peripheral and central hyperalgesia. Increasing evidence supports the use of brain-gut behavioral therapies, such as gut-directed hypnotherapy and cognitive behavior therapy, as effective treatments for a variety of DGBIs. However, the efficacy of neuromodulators or cognitive behavior therapy in treating esophageal DGBI and related symptoms remains largely unexplored. The primary objective of this study is to examine the efficacy of neuromodulators in managing esophageal DGBI. Additionally, we will explore various classes of neuromodulators and subtypes of esophageal DGBI to ascertain whether there are differing levels of effectiveness across these conditions. The findings from this study will contribute to a better understanding of the pathophysiology of esophageal DGBI and GERD with refractory symptoms. These clinical insights may then offer valuable guidance for future therapeutic approaches in DGBI patients who experience esophageal symptoms and do not respond to PPI treatment.

**Key words:** gastroesophageal reflux disease, disorders of gut-brain interaction, neuromodulators

## 7. Background and Objectives of the Research Project

( Please provide a detailed description of the background, objectives, significance of this research project, as well as the research status both domestically and internationally related to this project. Also, include a review of important references and literature. )

#### Research Background

#### ◆Pathophysiological Mechanisms and Importance of Gastroesophageal Reflux Disease (GERD)

Gastroesophageal reflux disease (GERD) is defined as a condition where stomach contents flow back into the esophagus, resulting in symptoms or mucosal injury. Common typical symptoms include heartburn or acid reflux, while atypical symptoms may include chest tightness, a sensation of a foreign body in the throat, hoarseness, or chronic cough. Clinically, GERD is a common chronic disease. In the United States, where symptoms occur at least once a week, up to 30% of adults are affected by GERD; in East Asia, the prevalence is 5-10%, but there is a growing trend in its incidence.

There are many possible pathogenic mechanisms for GERD, including lower esophageal sphincter (LES) dysfunction or structural abnormalities, ineffective esophageal motility, esophageal mucosal integrity defects, esophageal hypersensitivity, the formation of acid pockets after meals, the composition of gastric refluxate, and delayed gastric emptying. Currently, the most common diagnostic method involves observing damage to the distal esophageal mucosa through endoscopy or confirming abnormal gastric acid exposure via a 24-hour pH monitoring test. Based on the results of endoscopy and esophageal pH monitoring, GERD patients can be classified into two categories: erosive esophagitis (EE) and non-erosive reflux disease (NERD).

Repeated gastric acid exposure to the distal esophagus not only causes mucosal damage but may also lead to severe complications such as esophageal stricture, Barrett's esophagus, and esophageal adenocarcinoma. Statistics show that in the United States, medical and non-medical losses due to GERD exceed \$930 million annually. Therefore, GERD has become an important issue both clinically and in national public health policies in recent years.

#### **♦** Disorders of gut-brain axis interaction in esophagus

Disorders of gut-brain axis interaction (DGBI) refer to gastrointestinal diseases that present with symptoms but no organic abnormalities, which were previously referred to as functional gastrointestinal disorders. In the recent Rome IV criteria, <sup>11</sup> In the esophageal context, the Rome IV criteria define five conditions: functional chest pain, reflux hypersensitivity (RH), functional heartburn (FH), globus, and functional dysphagia. Epidemiologically, the prevalence of esophageal disorders related to gut-brain axis interaction is still not well understood. Past population-based

remains unclear to this day.

Further generation-based analysis of the population with psychogenic chest pain revealed that approximately 32-35% of them were diagnosed with functional chest pain. <sup>14</sup> In terms of reflux hypersensitivity, among patients with non-erosive mucosal damage in the esophagus, approximately 10-36% are diagnosed with esophageal hypersensitivity. <sup>15,16</sup> Functional heartburn has an unknown prevalence due to the limitations of current diagnostic tools and receiver operating characteristic (ROC) curves. Globus, on the other hand, is a commonly encountered disorder of gut-brain axis interaction in clinical practice. Research reports indicate that 46% of healthy adults have

experienced globus at some point.<sup>17</sup> Functional dysphagia is the least common, and its prevalence

In terms of definition, patients must have chronic esophageal symptoms lasting at least three months, with the first occurrence of symptoms being more than six months before the diagnosis of the disease. Additionally, structural, inflammatory, motility, and metabolic abnormalities in the esophagus must be excluded. Therefore, to diagnose esophageal disorders related to gut-brain axis interaction, upper gastrointestinal endoscopy, esophageal pH-impedance testing, and high-resolution esophageal manometry are required to exclude other esophageal diseases that may cause similar symptoms. Regarding the pathophysiological mechanisms, it is currently believed that they may be related to esophageal visceral hypersensitivity and hypervigilance, but the exact mechanisms still require further research for confirmation. In terms of diagnostic criteria, according to the Rome IV criteria, the definition is as follows:<sup>11</sup>

#### ➤ Functional Chest Pain:

- (1) Occurs ≥1 time per week with non-cardiac chest pain or chest tightness;
- (2) No associated heartburn or dysphagia;
- (3) Symptoms are not related to gastroesophageal reflux disease (GERD) or eosinophilic esophagitis;
- (4) No significant esophageal motility disorders.

#### > Functional Heartburn:

- (1) Occurs ≥2 times per week with substernal symptoms such as heartburn or chest pain;
- (2) Symptoms do not improve with antisecretory therapy;
- (3) Symptoms are not related to gastroesophageal reflux disease (GERD) or eosinophilic esophagitis;
- (4) No significant esophageal motility disorders.

#### > Reflux Hypersensitivity (Esophageal Hypersensitivity):

- (1) Occurs ≥2 times per week with substernal symptoms such as heartburn or chest pain;
- (2) Endoscopy is normal, and eosinophilic esophagitis must be excluded;
- (3) No significant esophageal motility disorders;

(4) Esophageal pH or pH-impedance testing shows normal acid exposure levels, but reflux is associated with symptoms.

#### **➢** Globus:

- (1) Occurs ≥1 time per week with persistent or intermittent, non-painful sensation of a lump in the throat, with no organic lesions confirmed through clinical examination, laryngoscopy, or endoscopy;
- (2) Symptoms occur between meals, with no dysphagia or odynophagia, and no gastric metaplasia in the proximal esophagus (gastric inlet patch);
- (3) Symptoms are not related to gastroesophageal reflux disease (GERD) or eosinophilic esophagitis;
- (4) No significant esophageal motility disorders.

#### > Functional Dysphagia:

- (1) Occurs ≥1 time per week with a sensation of obstruction or abnormal feeling when solids or liquids pass through the esophagus;
- (2) Symptoms are not related to esophageal mucosal or structural abnormalities;
- (3) Symptoms are not related to gastroesophageal reflux disease (GERD) or eosinophilic esophagitis;
- (4) No significant esophageal motility disorders.



Figure 1: Diagnostic Spectrum Classification of Gastroesophageal Reflux Disease (GERD) and Disorders of Gut-Brain Axis Interaction (DGBI).

# ◆ Physiological Tests for Diagnosing Gastroesophageal Reflux Disease (GERD) and Disorders of Gut-Brain Axis Interaction (DGBI)

The current diagnosis of gastroesophageal reflux disease (GERD) spectrum disorders is based on endoscopic examination, esophageal pH (or pH-impedance) testing results, and the association between reflux and symptoms. Among these, esophageal pH testing, specifically the acid exposure time (AET), is the most important pathophysiological parameter used to differentiate GERD from disorders of gut-brain axis interaction (DGBI).<sup>18</sup> The measurement method involves calculating the

percentage of time during a 24-hour monitoring period in which the distal esophageal pH value is less than 4. The Lyon Consensus on the diagnosis of gastroesophageal reflux disease (GERD) states that an acid exposure time (AET) of less than 4% is considered physiological reflux, while an AET greater than 6% is considered pathological reflux. Additionally, if the total number of reflux episodes in 24 hours is less than 40, it is considered normal, while more than 80 episodes is considered abnormal. The combination of parameters such as acid exposure time (AET), number of acid reflux episodes, number of acid reflux episodes lasting more than five minutes, and the longest reflux episode duration can be used to assess the severity of reflux. By combining esophageal pH testing with impedance values, it is possible to detect the direction of reflux, as well as the reflux of weakly acidic, alkaline fluids, or gases. During the detection period, patients are required to record all esophageal symptoms occurring during the esophageal pH-impedance testing. The physician will then compare these recorded symptoms with the reflux events documented by the pH-impedance monitor to calculate the association between reflux and symptoms (Symptom Association Probability, SAP, and Symptom Index, SI).<sup>21</sup>

Based on the above criteria for esophageal pH testing and endoscopic examination results, patients with esophageal reflux symptoms can be classified into erosive esophagitis, non-erosive reflux disease, esophageal hypersensitivity, and functional heartburn. Erosive esophagitis is characterized by visible mucosal damage at the distal esophagus during endoscopy; non-erosive reflux disease is identified by normal mucosa on endoscopy and pathological prolongation of the acid exposure time (AET) at the distal esophagus on esophageal pH testing; esophageal hypersensitivity presents with a normal AET, but the symptoms are associated with reflux events (refluxate may be acidic, weakly acidic, or weakly alkaline) as seen on pH-impedance testing; functional heartburn occurs when there are symptoms of gastroesophageal reflux disease, but both endoscopic examination and AET are normal. For disorders of gut-brain axis interaction, including functional chest pain, globus, and functional dysphagia, in addition to normal endoscopic and AET results, patients must not have significant esophageal motility disorders and must meet the diagnostic criteria related to esophageal symptoms, as well as the onset and duration of symptoms.

Current diagnostic tools, such as questionnaires, proton-pump inhibitor trials, and endoscopic examination, have low sensitivity and specificity for diagnosing gastroesophageal reflux disease (GERD). While esophageal pH (or pH-impedance) testing is considered the gold standard for diagnosing GERD, it can only detect and diagnose reflux events that occur during the test period. Among these, catheter-based esophageal pH testing is limited because it can only detect reflux activity during the 24-hour test period. Additionally, patients may experience discomfort from the catheter, which could lead to changes in their daily activities, thereby potentially affecting the diagnostic results to varying degrees. • <sup>22-23</sup> The 96-hour wireless capsule-based esophageal pH monitoring, compared to the 24-hour esophageal pH-impedance testing, not only avoids the

discomfort caused by the catheter but also extends the monitoring period to 96 hours. Previous studies have indicated that up to one-third of patients diagnosed with functional heartburn based on 24-hour esophageal pH-impedance testing had their diagnosis corrected to non-erosive reflux disease after undergoing 96-hour wireless capsule-based esophageal pH monitoring. However, the 24-hour esophageal pH-impedance testing can improve the probability of diagnosing or excluding gastroesophageal reflux disease (GERD) by calculating the mean nocturnal baseline impedance (MNBI). The mean nocturnal baseline impedance is derived by recording the 10-minute average impedance values during the patient's sleep at three one-hour intervals (1:00, 2:00, 3:00). Recent studies have indicated that the mean nocturnal baseline impedance is associated with mucosal integrity, acid exposure time, and reflux symptoms. Legal 25, 26

## **◆**The Treatment Dilemma of Refractory Gastroesophageal Reflux Disease and Esophageal Brain-Gut Axis Communication Disorders

Proton pump inhibitors (PPIs) are the primary medications used to treat gastroesophageal reflux disease. Although they are highly effective in improving typical heartburn symptoms in patients with erosive esophagitis , <sup>27-29</sup> However, their effectiveness in treating non-erosive gastroesophageal reflux disease (NERD) is less than ideal. According to statistics, up to 50% of patients treated with proton pump inhibitors (PPIs) for suspected reflux symptoms still experience persistent symptoms. <sup>1,30</sup> Studies have indicated that most gastroesophageal reflux disease (GERD) patients who are unresponsive to proton pump inhibitor (PPI) treatment have a normal acid exposure time (AET). <sup>32</sup> In patients with heartburn who remain unresponsive to high-dose proton pump inhibitor (PPI) treatment, more than 90% are diagnosed with esophageal hypersensitivity or functional heartburn. <sup>31,32</sup> In addition, patients with pathological reflux may also have concurrent esophageal brain-gut axis communication disorders. The complex pathophysiological mechanisms of gastroesophageal reflux disease (GERD) and the limited understanding of brain-gut interaction contribute to the poor treatment outcomes in such patients. Recent consensus suggests that non-reflux factors, such as altered perception or visceral hypersensitivity, may be associated with the refractory symptoms of the esophagus. <sup>33</sup>

## **◆**Treatment Strategies for Refractory Gastroesophageal Reflux Disease and Esophageal Brain-Gut Axis Communication Disorders

The treatment strategies for refractory gastroesophageal reflux disease (GERD) and esophageal brain-gut axis communication disorders remain unclear. Currently, it is believed that esophageal hypervigilance, anxiety, and autonomic arousal are the primary factors influencing the severity of symptoms and the response to reflux burden. The Esophageal Hypervigilance and Anxiety Scale

(EHAS) has been recently validated in studies as an effective tool for assessing esophageal hypersensitivity.<sup>34</sup> Therefore, it is considered a helpful tool in diagnosing esophageal brain-gut axis communication disorders. Neuromodulators are medications used clinically to treat these disorders. Previous research has shown that neuromodulators can effectively reduce symptoms in patients with irritable bowel syndrome (IBS) or functional dyspepsia by modulating visceral hypersensitivity through central and peripheral mechanisms.<sup>35,36</sup> Therefore, using neuromodulators to regulate visceral hypersensitivity and esophageal hypervigilance in esophageal brain-gut axis communication disorders is considered a feasible strategy. However, a systematic review of the literature shows that among the few available randomized controlled trials, the efficacy of neuromodulators in the various subtypes of esophageal brain-gut axis communication disorders is inconsistent.<sup>37</sup> Therefore, whether neuromodulators can be widely used in the treatment of these disorders still requires more supporting evidence.

### **Research Objectives**

The objectives of this study:

To explore the impact of neuromodulators on disorders related to abnormal communication in the esophageal-brain-gut axis.

Hypothesis:

- (1) Patients with disorders related to abnormal communication in the esophageal-brain-gut axis experience esophageal symptoms due to visceral hypersensitivity and heightened esophageal sensitivity, which affect their physical and mental health, sleep, and quality of life. Neuromodulators may alleviate symptoms and their associated impacts.
- (2) The effectiveness of neuromodulators may vary among patients with different subtypes of esophageal-brain-gut axis communication disorders.
- (3) The effectiveness of different neuromodulators may vary within the same subtype of esophageal-brain-gut axis communication disorders.

### 8. Research Methods, Procedures, and Execution Progress

- 1. Please describe in detail the research methods adopted in this project and the reasons for choosing them.
- 2. Potential challenges and solutions expected during the project.
- **3.** If this is a continuous project, please also attach the progress report from the previous year or primary data.

#### Research Method

#### **Participant**

This project is a multi-center study. we will recruit cases from five medical centers in Taiwan, including 210 cases from our hospital and 400 cases from other centers (120 cases each from Chengda Hospital, Kaohsiung Medical University Hospital, and E-Da Hospital, and 40 cases from Chung Shan Medical University Hospital). A total of 610 cases are expected to be recruited.

This study is expected to last for 2 years, with the study period ending on December 31, 2025. We intend to recruit participants with esophageal symptoms related to disorders of the gut-brain axis communication from the Gastroenterology outpatient clinics.

#### **Inclusion criteria for participants:**

- 1. Age between 18 and 75 years, with clear consciousness and willingness to sign the informed consent form.
- 2. Participants with chronic esophageal symptoms related to esophageal-brain-gut axis communication disorders (such as heartburn, acid reflux, sensation of a foreign body in the throat, difficulty swallowing, chest pain, and chest tightness).

#### **Exclusion criteria for participants:**

- 1. Esophageal stricture, or a history of esophageal, gastrointestinal, or throat surgery.
- 2. Structural esophageal diseases (e.g., diverticula, esophageal rings), infectious esophagitis, erosive esophagitis, eosinophilic esophagitis.
- 3. Non-erosive gastroesophageal reflux disease or significant esophageal motility disorders.
- 4. A history or current diagnosis of esophageal, gastrointestinal, or other organ malignancies.
- 5. Significant endocrine or rheumatic autoimmune diseases that may affect gastrointestinal motility.
- 6. Continuous use of medications that may affect esophageal motility (e.g., anticholinergics, morphine-like drugs, nitrates, calcium channel blockers) within the past month.
- 7. Use of antidepressants, selective serotonin reuptake inhibitors, or other psychiatric medications within the past three months.
- 8. Pregnant or breastfeeding women.
- 9. Individuals with mental disorders or those unable to cooperate.

- 10. Known allergy to tricyclic antidepressants.
- 11. Known allergy to selective serotonin reuptake inhibitors.
- 12. Known allergy to any component of proton pump inhibitors.

#### Research Design Flowchart



#### Steps to Follow

In this study, each participant will first complete a questionnaire, which includes the Gastroesophageal Reflux Disease Questionnaire (GERDQ, PROMIS GERD, DSI & GSS, RSI), the Brief Esophageal Dysphagia Questionnaire (BEDQ), the Esophageal Hypervigilance and Anxiety Scale (EHAS), the Visceral Sensitivity Index (VSI), the Sleep and Psychological Well-being Questionnaire (Pittsburgh Sleep Quality Index [PSQI], Taiwan Depression Questionnaire [TDQ], State-Trait Anxiety Inventory [STAI], Functional Dyspepsia [FD] Questionnaire, Irritable Bowel Syndrome [IBS] Questionnaire, and the Quality of Life Questionnaire [SF-12, North East Esophageal Quality of Life Scale, NEQOL]). The time to complete these questionnaires is approximately 20 to 30 minutes.

Afterwards, participants will be randomly assigned using a computer system to receive one of the following treatments for 12 weeks: a neuroregulator, the tricyclic antidepressant (TCA), or the selective serotonin reuptake inhibitor (SSRI), or a 12-week control treatment with a proton pump inhibitor (PPI). We plan to recruit 70 participants for each treatment group: TCA, SSRI, and PPI, with each participant having a 1/3 chance of being assigned to one of these groups.

The tricyclic antidepressant (TCA) will be administered as a 25 mg enteric-coated tablet of Amitriptyline (Ministry of Health and Welfare Drug Registration No. 047966), taken twice daily. The neuroregulator - selective serotonin reuptake inhibitor (SSRI) will be administered as a 50 mg

enteric-coated tablet of Sertraline (Ministry of Health and Welfare Drug Registration No. 021780), taken once daily. The control medication - proton pump inhibitor (PPI) will be administered as a 30 mg oral dissolving tablet of Pantoprazole (Ministry of Health and Welfare Drug Registration No. 024273), taken once daily.

After the 12-week treatment period, participants will complete the questionnaire again to finalize the study.

#### **Multicenter Communication and Coordination Method**

The hospital directors of the participating institutions and the principal investigator, Dr. Lei Wei-Yi, will communicate and coordinate via email and a Line group established for the project. The research data collected by each center will be managed and stored by the respective center's director. The hospital directors will assist in consolidating the research data from their institution, and the electronic data will be coded for identification. After the data is compiled, it will be sent back to the principal investigator. Additionally, the research physicians and staff at each participating center will have regular video conferences (every 2 months) to discuss and report on the progress of the study.

#### **Statistical Analysis**

All data will undergo normality testing using the Kolmogorov-Smirnov test. If continuous variables follow a normal distribution, they will be expressed as means and standard deviations; if not, they will be presented as medians and interquartile ranges.

For categorical variables, the Chi-square test or Fisher's exact test will be used for analysis. Continuous variables that are normally distributed will be analyzed using the unpaired t-test, while non-normally distributed continuous variables will be analyzed using the Mann-Whitney U test.

For comparisons involving more than three groups, if the data are normally distributed, an ANOVA with post hoc tests will be conducted. If the data are non-normally distributed, the Kruskal-Wallis test will be applied. A p-value of less than 0.05 will be considered statistically significant.

Statistical analyses will be performed using SPSS 19 for Windows (SPSS, Inc., Chicago, IL, USA).

#### Clinical Significance and Originality of This Study

The originality of this study lies in its use of visceral sensitivity, mind-body connection, esophageal hypersensitivity, anxiety questionnaires, and functional gastrointestinal questionnaires

to explore the effects of neuromodulators on diseases related to esophageal-brain-gut axis communication abnormalities. Patients with such conditions often experience more severe esophageal symptoms due to excessive visceral sensitivity and esophageal hypersensitivity. We will further compare the therapeutic effects of neuromodulators across different subtypes of esophageal-brain-gut axis communication abnormalities. Additionally, we will investigate the differences in treatment outcomes using various types of neuromodulators for these conditions.

## 9. Expected Work Items and Specific Outcomes

- (1) Please list the expected tasks to be completed within the execution period.
- (2) Expected contributions to academic research and other applied areas.
- (3) Expected training that participants will receive.

#### 1. Work items expected to be completed.

In this study, we will explore the effects of neuromodulators on diseases related to abnormalities in the esophageal-brain-gut axis communication. We will also compare the efficacy differences between different medications and between different subtypes of esophageal-brain-gut axis communication abnormalities.

## 2. The anticipated contributions to academic research, national development, and other applications.

- (1) The data obtained from this study will allow us to understand the role of visceral sensitivity and esophageal awareness in esophageal-brain-gut axis communication abnormalities and refractory gastroesophageal reflux disease. It will also help us establish the role of neuromodulators in esophageal-brain-gut axis communication abnormalities and their impact on the regulation of brain-gut axis communication.
- (2) Clinically, patients with esophageal-brain-gut axis communication abnormalities often experience delayed diagnoses and poor treatment outcomes. The results of this study will enable us to intervene early and accurately in such brain-gut axis communication abnormality cases, helping clinical healthcare providers develop precise and effective treatment strategies.

#### 3. The expected training for the participating staff.

In addition to receiving general research training (such as experimental design and execution, questionnaire creation and completion, result analysis and statistics, chart creation, oral presentations, writing papers, and the submission process), participants will also have the opportunity to learn more specialized research design and numerical analysis techniques.

#### 10. References

- 1. Delshad SD, Almario CV, Chey WD, et al. Prevalence of gastroesophageal reflux disease and proton pump inhibitor refractory symptoms. Gastroenterology 2020;158:1250–1261.e2.
- 2. Peery AF, Crockett SD, Barritt AS, et al. Burden of gastrointestinal, liver, and pancreatic diseases in the United States. Gastroenterology 2015;149:1731–1741.e3.
- 3. Eusebi LH, Ratnakumaran R, Yuan Y, et al. Global prevalence of, and risk factors for, gastro-oesophageal reflux symptoms: a meta-analysis. Gut 2018;67:430-440.
- 4. Dodds WJ, Dent J, Hogan WJ, et al. Mechanisms of gastroesophageal reflux in patients with reflux esophagitis. N Engl J Med 1982;307:1547-52.
- 5. Kahrilas PJ, Dodds WJ, Hogan WJ, et al. Esophageal peristaltic dysfunction in peptic esophagitis. Gastroenterology 1986;91:897-904.
- 6. McCallum RW, Berkowitz DM, Lerner E. Gastric emptying in patients with gastroesophageal reflux. Gastroenterology 1981;80:285-91.
- 7. Mitchell DR, Derakhshan MH, Robertson EV, et al. The role of the acid pocket in gastroesophageal reflux disease. J Clin Gastroenterol 2016;50:111-9.
- 8. Gyawali CP, Kahrilas PJ, Savarino E, et al. Modern diagnosis of GERD: the Lyon Consensus. Gut 2018;67:1351-1362.
- 9. Katzka DA, Pandolfino JE, Kahrilas PJ. Phenotypes of Gastroesophageal Reflux Disease: Where Rome, Lyon, and Montreal Meet. Clin Gastroenterol Hepatol 2020;18:767-776.
- 10. Francis DO, Rymer JA, Slaughter JC, et al. High economic burden of caring for patients with suspected extraesophageal reflux. Am J Gastroenterol 2013;108:905-11.
- 11. Drossman DA. Functional gastrointestinal disorders: history, pathophysiology, clinical features and Rome IV. Gastroenterology 2016;150:1262-1279, e2.
- 12. Locke GR 3rd, Talley NJ, Fett SL, et al. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology 1997;112:1448–1456.
- 13. Eslick GD, Jones MP, Talley NJ. Non-cardiac chest pain: prevalence, risk factors, impact and consulting—a population-based study. Aliment Pharmacol Ther 2003; 17:1115–1124.
- 14. Fass R, Dickman R. Non-cardiac chest pain: an update. Neurogastroenterol Motil 2006;18:408–417.
- 15. Kushnir VM, Sayuk GS, Gyawali CP. The effect of antisecretory therapy and study duration on ambulatory esophageal pH monitoring. Dig Dis Sci 2011; 56:1412–1419.
- 16. Savarino E, Zentilin P, Tutuian R, et al. Impedance-pH reflux patterns can differentiate non-erosive reflux disease from functional heartburn patients. J Gastroenterol 2012;47:159–168
- 17. Moloy PJ, Charter R. The globus symptom. Incidence, therapeutic response, and age and sex relationships. Arch Otolaryngol 1982;108:740–744.
- 18. Roman S, Gyawali CP, Savarino E, et al. Ambulatory reflux monitoring for diagnosis of gastro-esophageal reflux disease: Update of the Porto consensus and recommendations from an international consensus group. Neurogastroenterol Motil 2017;29:1-15.
- 19. Johnson LF, Demeester TR. Twenty-four-hour pH monitoring of the distal esophagus. A quantitative measure of gastroesophageal reflux. Am J Gastroenterol 1974;62:325-32.
- 20. Sifrim D, Castell D, Dent J, Kahrilas PJ. Gastro-oesophageal reflux monitoring: review and consensus report on detection and definitions of acid, non-acid, and gas reflux. Gut 2004;53:1024-31.
- 21. Ghillebert G, Janssens J, Vantrappen G, Nevens F, Piessens J. Ambulatory 24 hour intraoesophageal pH and pressure recordings v provocation tests in the diagnosis of chest pain of oesophageal origin. Gut 1990;31:738-44.
- 22. Kahrilas PJ, Shaheen NJ, Vaezi MF. American Gastroenterological Association Institute technical review on the management of gastroesophageal reflux disease. Gastroenterology 2008;135:1392-1413, 1413.e1-5.
- 23. Vaezi MF, Schroeder PL, Richter JE. Reproducibility of proximal probe pH parameters in 24-hour ambulatory esophageal pH monitoring. Am J Gastroenterol 1997;92:825-9.

- 24. Penagini R, Sweis R, Mauro A, et al. Inconsistency in the Diagnosis of Functional Heartburn: Usefulness of Prolonged Wireless pH Monitoring in Patients With Proton Pump Inhibitor Refractory Gastroesophageal Reflux Disease. J Neurogastroenterol Motil 2015;21:265-72.
- 25. Kandulski A, Weigt J, Caro C, et al. Esophageal intraluminal baseline impedance differentiates gastroesophageal reflux disease from functional heartburn. Clin Gastroenterol Hepatol 2015;13:1075-81.
- 26. Woodland P, Al-Zinaty M, Yazaki E, et al. In vivo evaluation of acid-induced changes in esophageal mucosa integrity and sensitivity in non-erosive reflux disease. Gut 2013;62:1256-61.
- 27. Chiba N, De Gara CJ, Wilkinson JM, et al. Speed of healing and symptom relief in grade II to IV gastroesophageal reflux disease: a meta-analysis. Gastroenterology 1997;112:1798-810.
- 28. Sabesin SM, Berlin RG, Humphries TJ, et al. Famotidine relieves symptoms of gastroesophageal reflux disease and heals erosions and ulcerations. Results of a multicenter, placebo-controlled, dose-ranging study. USA Merck Gastroesophageal Reflux Disease Study Group. Arch Intern Med 1991;151:2394-400.
- 29. Dean BB, Gano AD, Jr., Knight K, et al. Effectiveness of proton pump inhibitors in nonerosive reflux disease. Clin Gastroenterol Hepatol 2004;2:656-64.
- 30. El-Serag H, Becher A, Jones R. Systematic review: persistent reflux symptoms on proton pump inhibitor therapy in primary care and community studies. Aliment Pharmacol Ther. 2010;32(6):720–37.
- 31. Patel A, Sayuk GS, Gyawali CP. Prevalence, characteristics, and treatment outcomes of reflux hypersensitivity detected on pH-impedance monitoring. Neurogastroenterol Motil 2016;28:1382-1390.
- 32. Roman S, Keefer L, Imam H, et al. Majority of symptoms in esophageal reflux PPI non-responders are not related to reflux. Neurogastroenterol Motil 2015;27:1667-1674.
- 33. Aziz Q, Fass R, Gyawali CP, et al. Functional esophageal disorders. Gastroenterology. 2016;150:1368–79.
- 34. Taft TH, Triggs JR, Carlson DA, et al. Validation of the oesophageal hypervigilance and anxiety scale for chronic oesophageal disease. Aliment Pharmacol Ther 2018;47:1270-1277.
- 35. Ford AC, Talley NJ, Schoenfeld PS, et al. Efficacy of antidepressants and psychological therapies in irritable bowel syndrome: systematic review and meta-analysis. Gut. 2009;58(3):367-378.
- 36. Talley NJ, Ford AC. Functional dyspepsia. New England Journal of Medicine. 2015;373(19):1853-1863.
- 37. Weijenborg PW, de Schepper HS, Smout AJ, et al. Effects of antidepressants in patients with functional esophageal disorders or gastroesophageal reflux disease: a systematic review. Clin Gastroenterol Hepatol 2015;13(2):251-259.e251.